CLINICAL TRIAL: NCT06110884
Title: Effectiveness of Music Therapy for Speech Delay and Prosody Disorder in Children With Autism
Brief Title: Music Therapy for Speech and Prosody in Autistic Children (MTSPAC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202307099RIND
Record Dates: First submitted 2023-10-24; First posted 2023-11-01 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-09

CONDITIONS: Autism; Language Delay; Speech Disorders in Children
MeSH Terms: conditions — Autistic Disorder; Language Development Disorders | interventions — Music Therapy; Speech Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy group (Experimental)
  Interventions: Behavioral: music therapy, speech therapy
- Control group (Active Comparator)
  Interventions: Behavioral: speech therapy

INTERVENTIONS:
Behavioral: music therapy, speech therapy — receive group music therapy in addition to traditional language therapy
  Arms: Music therapy group
Behavioral: speech therapy — receive only traditional language therapy
  Arms: Control group

SUMMARY:
This research is a single-blind randomized controlled trial, where the investigators plan to recruit 40 children with autism, randomly divided into two groups. The music therapy intervention group will receive an hour of group music therapy in addition to traditional language therapy. The control group will receive only traditional language therapy. The trial will last for 8 weeks, and participants in both groups will be assessed before and after the trial.

During the study, the investigators will use professional recording equipment to record their speech and use the speech analysis software to objectively compare whether there are significant differences in prosody between the two groups of children with autism before and after the intervention. Besides the acoustic measurement the investigators also assess the language abilities autism trait performance, adaptive function, emotional behavior, and parent-child stress levels.

DETAILED DESCRIPTION:
This research is a single-blind randomized controlled trial, where the investigators plan to recruit 40 children with autism, randomly divided into two groups. The music therapy intervention group will receive an hour of group music therapy in addition to traditional language therapy. The control group will receive only traditional language therapy. The trial will last for 8 weeks, and participants in both groups will be assessed before and after the trial.

During the study, the investigators will use professional recording equipment to record their speech and use the speech analysis software to objectively compare whether there are significant differences in prosody between the two groups of children with autism before and after the intervention. Besides the acoustic measurement the investigators also assess the language abilities autism trait performance, adaptive function, emotional behavior, and parent-child stress levels.

The study hypothesizes that music therapy can contribute to improving language development delays in children with autism and may enhance their language development further by ameliorating prosody abnormalities. The investigators hope that this research can propose more diversified therapeutic methods for language development in children with autism.

ELIGIBILITY:
Inclusion Criteria:

* children with autism
* aged 3-5 y/o
* children with speech delay (T-score of Preschool Language Scale < 40)
* Mandarin as first language

Exclusion Criteria:

* children with other neurological diseases
* children without verbal output
* children with articulation or voice disorder

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Revised version of the Preschool Language Scale (PLS) | 8 weeks
  assess the language abilities of children, minimum value 0, maximum value 83, higher scores means a better outcome
Checklist for Autism Spectrum Disorder-Chinese Version (CASD-C) | 8 weeks
  evaluate autism trait performance

SECONDARY OUTCOMES:
Child Behavior Checklist for Ages 1½-5 (CBCL 1½-5) | 8 weeks
  evaluate emotional behavior
Parenting Stress Index | 8 weeks
  evaluate parent-child stress levels, minimum value 36, maximum value 180, higher scores means a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsin-chu branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No
We would like to consider sharing the acoustic measurement data with other researchers